CLINICAL TRIAL: NCT06987409
Title: Continuous Erector Spinae Block for Analgesia Following Lumbar Decompression: A Randomized Controlled Study
Brief Title: Continuous Erector Spinae Block for Analgesia Following Lumbar Decompression
Acronym: Lumbar-ESP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB 56541
Record Dates: First submitted 2024-08-23; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Spinal Stenosis; Lumbar Radiculopathy; Persistent Postsurgical Pain
Keywords: Erector spinae block; Regional anesthesia
MeSH Terms: conditions — Spinal Stenosis; Radiculopathy; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: In this trial, the investigators are investigating the efficacy of using a continuous erector spinae plane block that delivers Ropivacaine (compared to normal saline (placebo)) for managing post-operative pain following spine surgery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Nova Scotia Health (NSH) pharmacy will prepare either Ropivacaine or normal saline in identical elastomeric pumps labelled as "study drug" such that the patient, clinical staff and the researchers are blinded to assigned group. The pharmacy will maintain the assignment list, only unmasking assignment in cases of suspected local anesthetic systemic toxicity (LAST) or allergic reactions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector spinae plane catheter with Ropivacaine (Experimental): All study patients will have two catheters inserted during surgery (i.e. on either side of the spinal cord), but patients in this arm will receive Ropivacaine through the cathedars in addition to normal medications for post-operative pain.
  Interventions: Procedure: Continuous erector spinae plane block
- Erector spinae plane catheter with normal saline (Placebo Comparator): All study patients will have two catheters inserted during surgery (i.e. on either side of the spinal cord), but patients in this arm will receive normal saline (placebo) through the cathedars in addition to normal medications for post-operative pain.
  Interventions: Procedure: Continuous erector spinae plane block

INTERVENTIONS:
Procedure: Continuous erector spinae plane block — The attending surgeon or fellow will place the erector spinae plane catheters in the operating room. Following decompression +/- fusion of the lumbar spine, catheters will be placed under direct vision. The tips of the catheters will be placed superficial to the transverse processes, instrumentation, and bone graft of the lumbar spine, as applicable to the procedure. These will be deep to the erector spinae muscles, which will be closed on top of the catheters.

SUMMARY:
Lumbar spinal surgery is common, and the incidence of spinal fusion has increased dramatically over the past three decades. Patients requiring spinal surgery are typically prescribed several analgesics, (including opioids) while awaiting surgery. Postoperatively, use of high doses of opioids or anti-inflammatory medications have drawbacks. Severe post-operative pain is reported by 45-80% of patients and rates are generally higher in the opioid tolerant patients.

Regional anesthesia (blocking nerves with local anesthetics) works locally, thereby avoiding many side effects associated with other analgesics. One type of nerve block is called erector spinae plane block (ESP). Single injection nerve blocks have been found to decrease pain, nausea, and opioid consumption, while increasing patient satisfaction and quality of recovery. However, these effects only last for 24 hours or less while the worst pain occurs around 36 hours after surgery. Surgeon-placed indwelling catheters could allow infusions of local anesthetics for 54 hours.

This randomized control trial seeks to assess the effectiveness of surgeon-placed ESP catheters for pain control after lumbar spine surgery.

Hypothesis: Patients receiving a cESP will have less pain, improved quality of recovery, and opioid use following lumbar fusion surgery than those receiving current standard of care pain management.

Methodology: Adult patients undergoing lumbar spine surgery under orthopedic surgery in Halifax will be eligible. The study will include 100 participants, randomly assigned to 2 study arms of 50 participants (1:1 basis to Ropivacaine and placebo groups). At the end of surgery, the surgeon will place the ESP catheters in all study patients under sterile conditions before closing the wound. Ropivacaine 0.5% or normal saline (placebo) 15ml will be injected through each catheter (total 30ml). In the postanesthetic care unit (PACU), two elastomeric pumps will be attached to the ESP catheters. These will be filled with either Ropivacaine 0.2% or normal saline (placebo). The elastomeric pumps are small bottle that patients can carry with them after discharge home. The pumps automatically run at an infusion rate of 10 ml/hr for 54 hours. All patients will also receive the standard of care for pain management for this patient population, which is opioid based with acetaminophen. A quality of recovery (QoR-15) questionnaire will be completed at 72 hours post-operatively. Pain, catheter complication, and opioid use data will be gathered from the patient's charts at 24, 48, and 72 hours post-operatively. At 3- and 6-month follow-ups, patients will complete the Brief Pain Inventory questionnaire. We will analyze differences in pain and opioid consumption at 24, 48, and 72 hours, quality of recovery index scores at 72 hours, postoperative complication rates, and persistent pain at 3 and 6 months.

DETAILED DESCRIPTION:
Hypothesis Our hypothesis is that a continuous erector spinae plane block (cESP) is an effective postoperative analgesia for lumbar decompression and interbody fusion patients.

Primary Study Objective To compare pain scores as measured by numeric rating scale (NRS) at 24 hours between continuous erector spinae plane block (cESP) and standard of care with placebo following lumbar fusion surgery.

Main Study Objectives

1. To compare the quality of recovery (QoR-15) at 72 hours for patients with a cESP with ropivacaine versus placebo.
2. To compare cumulative opioid consumption (in oral morphine equivalents (OME)) between cESP and placebo groups.
3. To compare time to discharge from hospital between cESP and placebo groups.
4. To compare adverse events between cESP and placebo groups.
5. To compare persistent postsurgical pain (PSPP) at 3 months between cESP and placebo.

1. Research Plan Subject Selection, Inclusion/exclusion criteria This study will include patients undergoing lumbar decompression and lumbar interbody fusion surgery under orthopedic surgery at the QEII Health Sciences Center in Halifax, Nova Scotia.

Number of participants The study will include a maximum of 100 participants, randomly assigned to 2 study arms of 50 participants. If a participant withdraws from the study and inclusion of their data is not possible, another participant will be recruited to the same study group.

Randomization and concealment Patients who have consented to the study, will be randomly assigned into two groups at the time of the operation, once the procedure has started. A computer-generated random number will be assigned and tracked by the central pharmacy to randomize patients on a 1:1 basis to the Ropivacaine and placebo groups.

The Nova Scotia Health Authority (NSHA) pharmacy will prepare either Ropivacaine 0.2% (2mg/ml) or normal saline in identical elastomeric pumps labelled as "study drug" such that the patient, clinical staff and the researchers are blinded to assigned group.

ESP block procedure - Study Intervention The attending surgeon or fellow will place the erector spinae plane catheters in the operating room. Following decompression +/- fusion of the lumbar spine, two 18g multiholed catheters will be placed under direct vision. A 17g Tuohy needle will be used to tunnel the catheters such that the insertion points are separate from the wound. The tips of the catheters will be placed superficial to the transverse processes, instrumentation, and bone graft of the lumbar spine, as applicable to the procedure. These will be deep to the erector spinae muscles, which will be closed on top of the catheters. The catheters will be secured to the skin using liquid skin adhesive (Dermabond) and a specialized dressing (Epiguard). Local anesthetic will be administered via the catheters after the wound is closed but before the patient emerges from general anesthesia. Ropivacaine 0.5% or normal saline (placebo) 15ml will be injected through each catheter (total 30ml).

Postoperative care In the postanesthetic care unit (PACU), two elastomeric pumps will be attached to the ESP catheters. These will be filled with either Ropivacaine 0.2% or normal saline (placebo). The elastomeric pumps run at an infusion rate of 10ml/hr for 54 hours.

When the patients have met normal PACU discharge criteria they will be transferred to the orthopedics ward. The orthopedics team will determine when the patient is ready for discharge from hospital. Many patients are discharged the following day. If the study patients are discharged prior to the end of the infusion, they would take the elastomeric pump home with them to continue the infusion at home.

All patients in the study will have ESP catheters placed. Other than that, patients will receive all the usual pain medications they normally would in the postoperative period. Patients in the treatment group will be receiving an erector spinae plane block with ropivacaine in addition to usual pain management while patients in the control group will be receiving placebo (saline) via the erector spinae plane catheter in addition to usual pain management.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged >18 years) patients
* Undergoing lumbar decompression surgery +/- fusion
* Under the orthopedic surgery team

Exclusion Criteria:

* Surgery on an emergency basis (level 1, 2 or 3; <8 hours)
* An ejection fraction <30%
* Severe pre-existing liver disease (Child B or C)
* Severe kidney disease (Glomerular filtration rate (GFR) <30 (mL/min/1·73m²))
* An allergy to ropivacaine
* Weight <50 kg
* Unable to provide valid consent to study prior to surgery

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | 24 hours
  Patient rate pain level according to a numbered scale (0-10 with worse pain being rated higher).

SECONDARY OUTCOMES:
Quality of recovery (QoR-15) | 72 hours
  Questionnaire includes five domains of recovery after surgery: patient support, comfort, emotions, physical independence, and pain. Each item is graded on a eleven-point Likert scale with QoR-15 scores ranging from 0 (extremely poor quality of recovery) to 150 (excellent quality of recovery).
Cumulative opioid consumption (in oral morphine equivalents (OME)) | 72 hours
  Quantitative measure of opioid use to be recorded at 24, 48, and 72 hours.
Time to discharge from hospital | Up to 30 days
  Quantitative measure of the hours between surgery and discharge.
Adverse events | 30 days
  Includes recording of postoperative nausea and vomiting (PONV), pneumonia, respiratory failure, wound infection, sepsis, arrhythmias, readmission to hospital within 30 days, and hospital mortality.
Persistent postsurgical pain (PSPP) | 3 months and 6 months
  Based on the Brief Pain Inventory. Average pain in the prior 24 hours will be rated on a scale from 0-10 with worse pain being rated higher.

IPD SHARING:
Plan to Share IPD: No